CLINICAL TRIAL: NCT05554315
Title: Speckle Plethysmography Pulse Transit Time as a Marker of Blood Pressure Changes
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000849; 000849-CH
Record Dates: First submitted 2022-09-22; First posted 2022-09-26 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-08-28

CONDITIONS: Blood Pressure
Keywords: Optical Technique; Pulse Transit Time; Pearson Correlation Coefficient; Spg Waveform; Signal Quality; Natural History

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Male or female, aged 18 or greater in good general health as evidenced by medical history

SUMMARY:
Background:

Blood pressure is one of the key markers of cardiovascular health. High blood pressure, also called hypertension, can increase the risk of heart disease or stroke. Monitoring a person s blood pressure continuously over a 24-hour period at home is the best way to diagnose hypertension, but the equipment currently used to do it is cumbersome. This natural history study will test a new technique for monitoring blood pressure continuously over time.

Objective:

To test a new technique (speckle plethysmography) for measuring blood pressure in healthy adults.

Eligibility:

Healthy people aged 18 years and older.

Design:

Participants will come to the clinic a minimum of 2 times.

The screening visit will last up to 2 hours. Participants will have a physical exam. Their vital signs will be taken.

The clinical visit will last up to 1 hour. Participants will recline in a chair. Sensors to measure the activity of the heart will be placed on their chest. Different sensors will be placed on two fingers and one big toe. A device to measure blood pressure will be placed on one arm.

While wearing the sensors, participants will undergo 3 tests:

They will be asked to breathe slowly for 2 minutes.

They will be asked to solve a math problem.

They will immerse one hand or foot into an ice bath for up to 2 minutes.

Each test will be followed by a 5-minute recovery period.

Participants may elect to return for up to 3 more visits during the following week.

DETAILED DESCRIPTION:
Study Description:

This pilot study will investigate the use of a recently introduced optical technique, speckle plethysmography (SPG), as an alternative to photoplethysmography (PPG) for cuff-free blood pressure (BP) estimation using pulse transit time (PTT). Because of the increased signal quality of SPG in comparison to PPG, we hypothesize that pulse transit times calculated from ECG-SPG (sPTT) will have a better correlation to blood pressure than ECG-PPG (pPTT).

Objectives:

Primary Objective:

To examine the use of sPTT as a marker for blood pressure.

Secondary Objective:

To evaluate the use of sPTT in comparison to pPTT.

Exploratory Objectives:

1. To explore if the SPG waveform by itself can be used as a marker for blood pressure.
2. To evaluate signal quality of SPG in comparison to PPG across various skin tones.

Endpoints:

Primary Endpoints:

Pearson correlation coefficient between sPTT and BP.

Secondary Endpoints:

Pearson correlation coefficient between pPTT and BP.

Exploratory Endpoints:

1. Pearson correlation coefficient between BP and signal markers to be determined.
2. PPG Signal-to-noise ratio (SNR), SPG SNR

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Male or female, aged 18 or greater.
* In good general health as evidenced by medical history and physical.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Any active cardiovascular or pulmonary disorders or use of vasoactive medications.
* History of aneurysm or stroke.
* Pregnant by history.
* History of fainting or seizures.
* An open cut, sore, or bone fracture on or near the hands or feet.
* Known retinopathy, intraocular lens implantation, or glaucoma.
* Any other condition that in the opinion of the investigator would place the participant at unacceptable risk.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male or female, aged 18 or greater in good general health as evidenced by medical history
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2023-04-19 (Actual); Primary Completion 2025-08-05 (Actual); Study Completion 2025-08-08 (Actual)

PRIMARY OUTCOMES:
Use of sPTT as a marker for blood pressure. | 1 year
  To examine the use of sPTT as a marker for blood pressure.

SECONDARY OUTCOMES:
use of sPTT in comparison to pPTT | 1 year
  To evaluate the use of sPTT in comparison to pPTT.

CONTACTS AND LOCATIONS:
Overall Officials: Bruce J Tromberg, Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_000849-CH.html